CLINICAL TRIAL: NCT04590677
Title: Prediction of the Onset of Term and Preterm Labour (PREDICT)
Brief Title: Prediction of the Onset of Term and Preterm Labour
Acronym: PREDICT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: SPD Development Company Limited (Industry); Borne Charity (Unknown)
Responsible Party: Sponsor
Other Study IDs: C&W19/037
Record Dates: First submitted 2020-09-21; First posted 2020-10-19 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Preterm Pregnancy; Preterm Birth; Preterm Birth Complication; Preterm Premature Rupture of Membrane; Preterm Labor
Keywords: Preterm; Biomarker; Pregnancy
MeSH Terms: conditions — Premature Birth; Preterm Premature Rupture of the Membranes; Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood - Extraction for proteonomic and transcriptomic studies, single cell RNA extraction, DNA extraction and identification of biomarker.
  Urine - Metabolomic studies, single cell RNA, proteonomic and transcriptomic studies and identification of biomarker.
  Swabs - Cytokine analysis, microbiome Rectal swabs - cytokine and microbiome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Pregnant women at 36 weeks gestational age, who are not expected to have risk factors for preterm birth, n=150.
  Interventions: Other: Samples required from group 1 (procedure within observational study)
- Group 2: Pregnant women who have presented with signs and symptoms of threatened preterm labour (e.g. ruptured membranes, contractions, bleeding), at or after 24 weeks gestation, n=50.
  Interventions: Other: Samples required from group 2 (procedure within observational study)

INTERVENTIONS:
Other: Samples required from group 1 (procedure within observational study) — * Weekly maternal blood samples to be taken
  * Daily urine samples to be collected
  * One rectal swab at the initial visit only
  * Weekly vaginal swabs
  * Daily Heart rate monitoring (only applicable to a subset of women in group 1)
  Groups: Group 1
Other: Samples required from group 2 (procedure within observational study) — * Weekly maternal blood samples to be taken
  * Daily urine samples to be collected
  * One rectal swab at the initial visit only
  * Weekly vaginal swabs
  Groups: Group 2

SUMMARY:
This study will collect samples from pregnant women in order to identify biomarkers that relate to onset of spontaneous preterm labour.

DETAILED DESCRIPTION:
Preterm birth is not a single entity but rather multifactorial The mechanisms underlying preterm birth are multifactorial and include stretch, oxidative stress, inflammation, infection and thrombosis. 85% of women have no identifiable risk factors for preterm birth and there is a requirement to develop a biomarker which can be used early in pregnancy to identify such women at risk. Equally important is to have a detection tool which will allow us to offer an individualised approach to preterm birth prevention and the women to benefit personalised surveillance and timely preventative measures such as cervical cerclage or progesterone.

The aim of this study is to collect samples from pregnant women in order to identify biomarkers that relate to onset of spontaneous preterm labour. We will use maternal blood, urine and vaginal secretion to look for biomarkers in these samples which can be use in the clinical setting to determine which women will go on to give birth preterm. This will allow clinicians to correctly identify these women and initiate treatment in the right woman to prevent preterm labour and birth. Equally important it will reduce unnecessary intervention and admission in those women who are not at risk.

ELIGIBILITY:
Group 1 inclusion criteria

* Pregnant woman
* 36 weeks gestational age

Group 1 exclusion criteria

* Risk factors for preterm birth (previous preterm birth or second trimester loss, cervical suture, previous cervical treatment, previous full dilatation caesarean, transabdominal suture).
* Planned Caesarean Section
* Any high-risk pregnancy conditions such as PET (pre-eclamptic toxaemia), OC (Obstetric cholestasis), FGR (fetal growth restriction)
* Unable to read written English
* Unable to provide informed consent
* Poor attendance with antenatal care
* Uncertain gestational age

Exclusion criteria for subset within group 1 using heart rate monitor

* Does not have access to an Apple iPhone or iPad with Bluetooth 4.0 (or later) and iOS 10.0 (or later)
* Skin condition where there is sensitivity to wearing a skin monitor
* Known heart condition or use of a pacemaker
* Taking any medications that may affect heart rate

Group 2 inclusion criteria

* Pregnant woman
* Presenting at or after 24 weeks gestational age and before 36 weeks / Symptoms of threatened preterm labour (abdominal pain) with fetal fibronectin level ≥ 50 ng/mL and without rupture of membranes
* In-utero transfer with suspected threatened preterm labour with evidence of cervical shortening and dilatation with or without a fetal fibronectin
* Rupture of membranes with or without contractions

Group 2 exclusion criteria

* Any high-risk pregnancy conditions such as PET (pre-eclampsia), OC (Obstetric cholestasis), FGR (fetal growth restriction)
* Unable to read written English
* Unable to provide informed consent
* Poor compliance with antenatal care
* Uncertain gestational age

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Relative change in biomarker concentration with respect to gestational age of onset of term and preterm labour | Group 1 from 36 weeks until delivery (approximately 6 weeks). Group 2 from admission at or beyond 24 weeks gestation until 42 weeks of gestation if not delivered.
  To use a combination of maternal blood, urine, rectal and vaginal swabs from pregnant to develop a biomarker to allow prediction of women at risk of preterm birth.

SECONDARY OUTCOMES:
Optimal thresholds for each biomarker and estimated associated sensitivity, specificity of each biomarker | Group 1 from 36 weeks until delivery (approximately 6 weeks). Group 2 from admission at or beyond 24 weeks gestation until 42 weeks of gestation if not delivered.
  * To determine the temporal relationship between concentration of each biomarker e.g. hCG (IU/L), Progesterone (µg/ml) and onset of labour.
  * For biomarkers that demonstrate a clinically relevant relationship with onset of labour e.g. hCG (IU/L), Progesterone (µg/ml), the clinical utility of the biomarker will be determined.
Correlation between the percentage of patients with reported demographic variables, lifestyle variables and clinical symptoms | Group 1 from 36 weeks until delivery (approximately 6 weeks). Group 2 from admission at or beyond 24 weeks gestation until 42 weeks of gestation if not delivered.
  To determine the correlation between the percentage of patients with reported demographic variables, lifestyle variables and clinical symptoms reported through questionnaires and a daily diary and the onset of preterm birth.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Singh, MRCOG, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngo TTM, Moufarrej MN, Rasmussen MH, Camunas-Soler J, Pan W, Okamoto J, Neff NF, Liu K, Wong RJ, Downes K, Tibshirani R, Shaw GM, Skotte L, Stevenson DK, Biggio JR, Elovitz MA, Melbye M, Quake SR. Noninvasive blood tests for fetal development predict gestational age and preterm delivery. Science. 2018 Jun 8;360(6393):1133-1136. doi: 10.1126/science.aar3819. PMID 29880692
- [Background] Heng YJ, Di Quinzio MK, Permezel M, Rice GE, Georgiou HM. Interleukin-1 receptor antagonist in human cervicovaginal fluid in term pregnancy and labor. Am J Obstet Gynecol. 2008 Dec;199(6):656.e1-7. doi: 10.1016/j.ajog.2008.06.011. Epub 2008 Jul 21. PMID 18640661
- [Background] Heng YJ, Di Quinzio MK, Permezel M, Rice GE, Georgiou HM. Cystatin A protease inhibitor and cysteine proteases in human cervicovaginal fluid in term pregnancy and labor. Am J Obstet Gynecol. 2011 Mar;204(3):254.e1-7. doi: 10.1016/j.ajog.2010.10.912. Epub 2010 Dec 16. PMID 21167469